CLINICAL TRIAL: NCT05264077
Title: Efficacy of Dexmedetomidine Versus Midazolam for Early Extubation in Critically Ill Agitated Patients Undergoing Weaning
Brief Title: Efficacy of Dexmedetomidine vs Midazolam for Early Extubation in Critically Ill Agitated Patients Undergoing Weaning
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Momal Jaleel Khan, Dr.Momal jaleel khan, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MJKhan
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Agitation, Emergence
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): Inj.Dexmedetomidine(precidex ) 200mcg/2ml Given to participants in infusion form for 24 hours
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Midazolam (Experimental): Inj.midazolam 5mg/ml given to participants in infusion form for 24 hrs
  Interventions: Drug: Dexmedetomidine Hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Inj dexmedetomidine and inj midazolam given to two groups of participants and effects of both drugs will be observed for 24 hrs
  Other Names: Midazolam

SUMMARY:
Comparison of effect of dexmedetomidine and midazolam in icu patients who put on mechanical ventilation and show agitation on weaning.Selection of better agent minimises the drug related side effects like respiratory depression but also helps in weaning for early extubation,give hemodynamic stability and reduce morbidity and mortality in icu..

ELIGIBILITY:
Inclusion Criteria:

* all patients with age <60 irrespective of gendre

Exclusion Criteria:

- Patients who refuse to give consent, severely altered conscious level (GCS < 8/15), traumatic injury causing hypoxemia e.g., severe head / chest / facial trauma or pneumothorax, severe pneumonia, arrhythmia, impaired hearing or blindness, severe hepatic or renal disease, on neuromuscular blocking agents, recent myocardial infarction, use of anti-psychotics, hypersensitivity to any of the drug under study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Effective sedation in icu patients lead to successful 1weaning in icu patients | Upto 48 hrs
  Assess patients by using ramsay sedation score (score 1 =awake upto score 6=no response)

IPD SHARING:
Plan to Share IPD: No